CLINICAL TRIAL: NCT02304250
Title: The Effect of Dexamethasone on Safety of Thyroid Surgery
Brief Title: Dexamethasone and Wound Healing After Thyroid Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quanhong Zhou (Other)
Responsible Party: Sponsor-Investigator, Quanhong Zhou, Doctor, Shanghai 6th People's Hospital
Organization: Shanghai 6th People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2014-50
Record Dates: First submitted 2014-11-19; First posted 2014-12-01 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Wound Infection
MeSH Terms: conditions — Wound Infection | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group D (Active Comparator): Group D: dexamethasone group
  Interventions: Drug: Dexamethasone
- Group S (Placebo Comparator): Group S: saline group
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Dexamethasone — dexamethasone 1ml (5mg)
  Arms: Group D
Drug: saline — saline 1ml
  Arms: Group S

SUMMARY:
Dexamethasone is a potent glucocorticoid with analgesic and anti-emetic effects [1-3]. Perioperative single-dose dexamethasone therapy has been used for several purposes: to reduce post-operative nausea and vomiting (PONV), pain and sore throat. There are also some reports on beneficial effects of less cardiac arrhythmia, improved appetite and less edema from glucocorticoids. Preoperative small dose of dexamethasone was reported to prevent reversal laryngeal nerve injury and improve voice quality after thyroid surgery. While accepted wildly in clinical anesthesia practice, the immune-press related potential risks of side effects associated with dexamethasone, such as delayed wound healing, infection, as well as effects on blood sugar, make the use of perioperative single dose of glucocorticoid controversial. The effect of perioperative dexamethasone on wound healing varied with different types of surgery. The present study will observe the effect of dexamethasone on the safety of thyroid surgery.

DETAILED DESCRIPTION:
Patients who has the thyroid surgery for their thyroid cancer will be randomly allocated into two groups, either dexamethasone group or saline group. In the dexamethasone group, patients will receive 5mg dexamethasone iv right after general anesthesia induction while in the saline group, patients will have 1ml saline iv. The drainage fluid will be collected at 6 hours after surgery and on every morning after operation till the drainage tube is taken out. The total amount of drainage fluid and blood stain area in dressing will be collected and calculated after the operation. The C-reaction protein is checked in drainage fluid and in blood after operation. Besides, the pain scores of incision pain and throat pain will be evaluated. Postoperative nausea and vomit will be checked as well.

ELIGIBILITY:
Inclusion Criteria:

* Elective total thyroidectomy or hemithyroidectomy with lymphadenectomy for thyroid cancer

Exclusion Criteria:

* Age > 65 years, < 18 years
* Thyroid tumor with Grave's disease
* Thyroid tumor size over 5 cm
* Second or more than 2 times for thyroid surgery
* Non-traditional pathway for thyroid surgery
* ASA > II
* Pharyngitis
* Smoking, alcohol drinking history
* Contraindication or long term use of dexamethasone (allege, ulcer bleeding history, et al)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2013-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
the total wound drain after the operation, including the drain in bulb and stain area in dressings, | from postoperative day 0 to postoperative day 4

SECONDARY OUTCOMES:
patient pain scores, including incision pain and throat pain, | from postoperative day 0 to one month after operation
c-reaction protein levels in drainage fluid and blood during perioperative period. | from postoperative day 0 to postoperative day 4

OTHER OUTCOMES:
patient nausea/vomiting scores | from postoperative day 0 to 3 days after operation
other side effects from the surgery | from postoperative day 0 to one month after the operation

CONTACTS AND LOCATIONS:
Overall Officials: WEIPING JIA, Ph.D, Study Chair — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai 6Th People'S Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang H, Lu J, Wu Q, Wu B, Xu C, Fan Y, Zhou Q. A Perioperative Small Dose of Dexamethasone Enhances Postoperative Recovery by Reducing Volume and Inflammatory Contents in Wound Drainage After Thyroid Surgery: A Double-Blinded, Randomized, Prospective Study. World J Surg. 2019 Jul;43(7):1721-1727. doi: 10.1007/s00268-019-04986-0. PMID 30963205